CLINICAL TRIAL: NCT06891651
Title: Clinical Cohort Study of 21-gene Assay in Predicting the Prognosis of Elder Luminal-A Breast Cancer Patients With Axillary Lymph Node Metastasis
Brief Title: 21-gene in Elder Breast Cancer Patients With Lymph Node Metastasis
Acronym: QiluElderHope
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202407-026-1; 26010112002346 (Other Grant/Funding Number: Amoy Diagnostics Co., Ltd.)
Record Dates: First submitted 2025-02-21; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Metastatic; Breast Cancer Survival
Keywords: Breast cancer; 21-gene assay; Axillary lymph node metastasis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 21-gene assay in elder breast cancer with axillary lymph node metastasis: 21-gene assay will be performed not only in primary cancer site in breast but also in metastatic lymph nodes.

SUMMARY:
This study is a single-center, bidirectional cohort study. It aims to include 35 elderly (≥65 years old) Luminal A type breast cancer patients with axillary lymph node metastasis after surgery as the research subjects. After signing the informed consent, the patients who meet the inclusion criteria will have their various clinical and pathological data collected (preoperative imaging examinations, clinical and pathological information of the patients, basic disease conditions and medication strategies, surgical records, postoperative planned treatment plans and actual treatment situations, etc.), and their real adjuvant treatment situations (whether chemotherapy, radiotherapy, endocrine therapy, targeted therapy, etc. were performed after surgery) will be followed up and recorded. At the same time, paraffin tissues of breast cancer and metastatic lymph nodes of the patients will be collected from the pathology department of our hospital for 21-gene assay, and the recurrence risk index of the primary lesion and metastatic lymph nodes will be obtained using the risk index calculation logic of Amoy Diagnostics Company. An assessment will be conducted every 12 months after surgery until disease recurrence. After disease recurrence, survival follow-up will be conducted every three months until the patient's death. The predictive value of 21-gene assay for patient survival and whether chemotherapy is beneficial will be evaluated based on the follow-up data of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent；
* Female, age ≥ 65 years old；
* Patients who have undergone radical surgery for breast cancer (radical surgery refers to modified radical mastectomy, radical mastectomy or simple mastectomy + axillary lymph node dissection), and have been histologically confirmed to have axillary lymph node metastasis after surgery；
* Postoperative immunohistochemical typing and pTNM staging meet the following criteria:

  1. Luminal A type (ER and PR positive with a positive rate ≥ 20%, Her-2 gene negative, Ki67 < 15%), with pTNM staging of pTanyNanyM0.
  2. Or Luminal B, Her-2 gene negative type, with ER and PR positive and a positive rate ≥ 20%, Ki67 ≤ 30%, and pTNM staging of pTanyN1M0.
  3. Or age ≥ 70 years old, Luminal B, Her-2 gene negative type, with ER and PR positive and a positive rate ≥ 20%, Ki67 ≤ 30%, and pTNM staging of pTanyNanyM0.
  4. Or age ≥ 70 years old, but refuse or are unable to tolerate chemotherapy treatment, ER or PR positive, with pTNM staging of pTanyNanyM0；
* ECOG score 0-1；
* Expected survival time > 6 months.

Exclusion Criteria:

* Patients who have received preoperative neoadjuvant therapy in the past;
* Patients with bilateral breast cancer;
* Patients whose paraffin tissue specimens have been stored for more than 3 years at the start of the project;
* Patients with mental disorders who are unable to cooperate with subsequent treatment and follow-up;
* Patients with a history or evidence of disease, treatment or abnormal laboratory test values that may interfere with the trial results or prevent full participation in the study, or other situations deemed unsuitable for inclusion by the researcher, or those considered to have other potential risks and thus not suitable for participation in this study.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Qilu hospital of Shandong University or its medical alliance hospital
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether elderly Luminal-A breast cancer patients with axillary lymph node metastasis could benefit from 21-gene assay. | From enrollment to 80 years old（Average life expectancy）or mortality.
  All analyses will be conducted using SPSS 22.0. Comparisons between groups will be reported with 95% confidence intervals and p-values. Continuous variables will be presented as mean ± SD or median (min, max) based on distribution normality. Categorical variables will be described using frequencies (%).
  Disease-Free Survival (DFS) Unit of measure: Months from postoperative baseline Assessment: Time to first radiological recurrence (RECIST v1.1) or death Method: Kaplan-Meier analysis with log-rank test

SECONDARY OUTCOMES:
Whether elderly Luminal-A breast cancer patients with axillary lymph node metastasis could benefit from 21-gene assay | From enrollment to 80 years old（Average life expectancy）or mortality.
  Overall Survival (OS) Unit of measure: Months from enrollment Assessment: Time to all-cause mortality Method: Kaplan-Meier analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Zhu, M.D. & Ph.D., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertagnolli MM, Singh H. Treatment of Older Adults with Cancer - Addressing Gaps in Evidence. N Engl J Med. 2021 Sep 16;385(12):1062-1065. doi: 10.1056/NEJMp2106089. Epub 2021 Sep 11. No abstract available. PMID 34506087
- [Background] Lin J, Guo Z, Wang S, Zheng X. Omission of Chemotherapy in HR+/HER2- Early Invasive Breast Cancer Based on Combined 6-IHC Score? Clin Breast Cancer. 2021 Oct;21(5):e565-e574. doi: 10.1016/j.clbc.2021.01.011. Epub 2021 Jan 23. PMID 33674187
- [Background] Sparano JA, Gray RJ, Makower DF, Pritchard KI, Albain KS, Hayes DF, Geyer CE Jr, Dees EC, Goetz MP, Olson JA Jr, Lively T, Badve SS, Saphner TJ, Wagner LI, Whelan TJ, Ellis MJ, Paik S, Wood WC, Ravdin PM, Keane MM, Gomez Moreno HL, Reddy PS, Goggins TF, Mayer IA, Brufsky AM, Toppmeyer DL, Kaklamani VG, Berenberg JL, Abrams J, Sledge GW Jr. Adjuvant Chemotherapy Guided by a 21-Gene Expression Assay in Breast Cancer. N Engl J Med. 2018 Jul 12;379(2):111-121. doi: 10.1056/NEJMoa1804710. Epub 2018 Jun 3. PMID 29860917
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204